CLINICAL TRIAL: NCT04374149
Title: Interventional Study to Evaluate the Efficacy of Therapeutic Plasma Exchange (TPE) Alone or in Combination With Ruxolitinib in COVID-19 Positive Patients With PENN Grade 2, 3, 4 Cytokine Released Syndrome (CRS)
Brief Title: Therapeutic Plasma Exchange Alone or in Combination With Ruxolitinib in COVID-19 Associated CRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHU COVID-19-001
Record Dates: First submitted 2020-04-20; First posted 2020-05-05 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Cytokine Release Syndrome; COVID19
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19 | interventions — Plasma Exchange; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 - TPE Alone (Experimental): TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy
  Interventions: Procedure: Therapeutic Plasma Exchange
- 2 - TPE Plus Ruxolitinib (Experimental): TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy combined with ruxolitinib 5mg po twice daily (BID) beginning day prior to first TPE and continuing BID for total of 14 days.
  Interventions: Procedure: Therapeutic Plasma Exchange; Drug: Ruxolitinib

INTERVENTIONS:
Procedure: Therapeutic Plasma Exchange — TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy
Drug: Ruxolitinib — TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy combined with ruxolitinib 5mg po BID beginning day prior to first TPE and continuing BID for total of 14 days.
  Other Names: Therapeutic Plasma Exchange
  Arms: 2 - TPE Plus Ruxolitinib

SUMMARY:
This protocol will evaluate the efficacy of Therapeutic Plasma Exchange (TPE) alone or in combination with ruxolitinib in COVID positive patients with PENN grade 2, 3, 4 cytokine release syndrome (CRS). It is hypothesized that dual intervention of acute apheretic depletion of cytokines and concomitant suppression of production will produce superior amelioration of the cytokine load and to help to prevent cytokine load rebound. This protocol is envisioned as a pilot study (n=20) for hypothesis generation for future investigation.

DETAILED DESCRIPTION:
A virally mediated pandemic of 2020 is linked to a novel Beta Coronavirus (COVID-19) sharing subgenus classification with the severe acute respiratory syndrome (SARS) virus. The predominant modes of transmission are respiratory aerosolization and contaminated surface contact. COVID-19 infection is characterized by a wide range of severity and disease manifestations from asymptomatic to respiratory and multi organ failure. Definitive treatment is lacking, but there is an increasing awareness of its associated systemic cascade of inflammatory molecules that offers avenues to explore therapeutically.

Therapeutic plasma exchange (TPE) offers an immediate and scientifically grounded intervention for the removal of a host of pathogenic antibodies and toxic molecules by centrifugal separation of plasma or plasma membrane filtration. TPE in conjunction with Tocilizumab and steroids has been used successfully in the management of severe cytokine release syndrome (CRS) following chimeric antigen receptor T-cell therapy (CAR-T).

Precedence for consideration of TPE in a variety of inflammatory dominant disease states is also well known. Interest in adjuvant treatment for management of sepsis and multi organ dysfunction has been studied. TPE has also been used in three pediatric patients with pH1N1 influenza A acute respiratory failure and hemodynamic shock despite failure of best supportive care. All three survived with "good functional recovery."

Ruxolitinib is a Janus kinase (JAK) and signal transducer and activator of transcription (STAT) (JAK/STAT) pathway inhibitor which is FDA approved for polycythemia rubra vera, myelofibrosis and graft versus host disease. A murine model of CRS following CAR-T cellular therapy has been developed showing marked elevation of interleukin-6 (IL-6), interferon-gamma, tumor necrosis factor (TNF) alpha mimicking human CAR-T therapy induced CRS. Ruxolitinib treated mice demonstrated clinical amelioration and decrement in inflammatory cytokines. Incyte Corporation has announced plans to launch a Phase III trial of single agent ruxolitinib for COVID-19 associated cytokine storm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients positive for COVID-19 by polymerase chain reaction (PCR) assay or alternative accepted methodology
2. PENN class 2,3,4 CRS
3. Respiratory insufficiency with supplemental oxygen to maintain O2 sat greater than 89%
4. Clinically positive imaging by chest x-ray (CXR) or CT scan with evidence of bilateral pulmonary infiltrates, ground glass opacification or other pattern of consolidation felt likely to be linked to COVID infection or complication thereof
5. Age 12-80 years of age

Exclusion Criteria:

1. Pregnancy
2. Breast feeding
3. Class 3-4 New York Heart Association (NYHA) heart failure
4. Current use of synthetic disease modifying anti-rheumatic drugs (DMARDS) or IL-6 inhibitors or other immunosuppressive therapies outside of number five below
5. Current use of chronic corticosteroids if in excess of prednisone 10mg per day or equivalent
6. Suspected or confirmed clinically significant bacterial infection
7. History of tuberculosis (TB)
8. History of HIV
9. History of irritable bowel disease (IBD)
10. JAK inhibitor use within last 30 days
11. Creatinine clearance less than 15 ml / min
12. Absolute neutrophil count < 1000
13. Platelet count < 50,000
14. Clinical assessment that the trial could pose unacceptable risk by study participation
15. Current enrollment on another investigational protocol for COVID-19 induced CRS
16. Stage 4 obstructive lung disease with chronic hypoxic respiratory failure requiring supplemental O2 at baseline, or interstitial lung disease (ILD) with chronic hypoxic respiratory failure requiring supplemental O2 at baseline

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Larry Gluck, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant date (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available April 2021 through December 2021
Access Criteria: Data can be requested from the Principal Investigator via email and should include a description of the request and the associated project or use of the data.

REFERENCES:
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Jernigan DB; CDC COVID-19 Response Team. Update: Public Health Response to the Coronavirus Disease 2019 Outbreak - United States, February 24, 2020. MMWR Morb Mortal Wkly Rep. 2020 Feb 28;69(8):216-219. doi: 10.15585/mmwr.mm6908e1. PMID 32106216
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Xiao X, He X, Li Q, Zhang H, Meng J, Jiang Y, Deng Q, Zhao M. Plasma Exchange Can Be an Alternative Therapeutic Modality for Severe Cytokine Release Syndrome after Chimeric Antigen Receptor-T Cell Infusion: A Case Report. Clin Cancer Res. 2019 Jan 1;25(1):29-34. doi: 10.1158/1078-0432.CCR-18-1379. Epub 2018 Oct 15. PMID 30322878
- [Background] Busund R, Koukline V, Utrobin U, Nedashkovsky E. Plasmapheresis in severe sepsis and septic shock: a prospective, randomised, controlled trial. Intensive Care Med. 2002 Oct;28(10):1434-9. doi: 10.1007/s00134-002-1410-7. Epub 2002 Jul 23. PMID 12373468
- [Background] Rimmer E, Houston BL, Kumar A, Abou-Setta AM, Friesen C, Marshall JC, Rock G, Turgeon AF, Cook DJ, Houston DS, Zarychanski R. The efficacy and safety of plasma exchange in patients with sepsis and septic shock: a systematic review and meta-analysis. Crit Care. 2014 Dec 20;18(6):699. doi: 10.1186/s13054-014-0699-2. PMID 25527094
- [Background] Patel P, Nandwani V, Vanchiere J, Conrad SA, Scott LK. Use of therapeutic plasma exchange as a rescue therapy in 2009 pH1N1 influenza A--an associated respiratory failure and hemodynamic shock. Pediatr Crit Care Med. 2011 Mar;12(2):e87-9. doi: 10.1097/PCC.0b013e3181e2a569. PMID 20453703
- [Background] Porter D, Frey N, Wood PA, Weng Y, Grupp SA. Grading of cytokine release syndrome associated with the CAR T cell therapy tisagenlecleucel. J Hematol Oncol. 2018 Mar 2;11(1):35. doi: 10.1186/s13045-018-0571-y. PMID 29499750
- [Derived] Gluck WL, Callahan SP, Brevetta RA, Stenbit AE, Smith WM, Martin JC, Blenda AV, Arce S, Edenfield WJ. Efficacy of therapeutic plasma exchange in the treatment of penn class 3 and 4 cytokine release syndrome complicating COVID-19. Respir Med. 2020 Dec;175:106188. doi: 10.1016/j.rmed.2020.106188. Epub 2020 Nov 7. PMID 33190086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were hospitalized at the time of enrollment. They were identified and referred by the critical care service physicians.
Pre-assignment Details: Eligible patients were consecutively enrolled with the first 10 to cohort 1A and the second 10 to cohort 1B.
Groups:
- 1 - TPE Alone: Therapeutic Plasma Exchange (TPE), five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy
  Therapeutic Plasma Exchange: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy
- 2 - TPE Plus Ruxolitinib: Therapeutic Plasma Exchange (TPE), five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy combined with ruxolitinib 5mg po twice daily (BID) beginning day prior to first TPE and continuing BID for total of 14 days.
  Therapeutic Plasma Exchange: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or fresh frozen plasma (FFP) replacement if underlying coagulopathy
  Ruxolitinib: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy combined with ruxolitinib 5mg po twice daily (BID) beginning day prior to first TPE and continuing BID for total of 14 days.
Period: Overall Study
Arm/Group | 1 - TPE Alone | 2 - TPE Plus Ruxolitinib
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 - TPE Alone: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy
  Therapeutic Plasma Exchange: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy
- 2 - TPE Plus Ruxolitinib: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy combined with ruxolitinib 5mg po BID beginning day prior to first TPE and continuing BID for total of 14 days.
  Therapeutic Plasma Exchange: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy
  Ruxolitinib: TPE, five single plasma volume exchanges over 7 days (every day x 2 then every other day x 3) with albumin or FFP replacement if underlying coagulopathy combined with ruxolitinib 5mg po BID beginning day prior to first TPE and continuing BID for total of 14 days.
- Total: Total of all reporting groups
Arm/Group | 1 - TPE Alone | 2 - TPE Plus Ruxolitinib | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (12.6) | 57.4 (8.8) | 54.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 3 | 9 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 6 | 2 | 8
  White | 2 | 6 | 8
  Asian | 1 | 0 | 1
  Black | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 34.4 (10.2) | 36.0 (5.6) | 35.2 (7.9)
Days from COVID positive test to first therapeutic plasma exchange (TPE) [Median (Inter-Quartile Range); unit: Days] | 4.5 [3 to 6] | 9 [4 to 12] | 6.75 [3 to 12]
ABO Blood Group [Count of Participants; unit: Participants]
  A- | 1 | 1 | 2
  A+ | 2 | 2 | 4
  B+ | 2 | 1 | 3
  O+ | 5 | 6 | 11
Respiratory Status per Penn Class [Count of Participants; unit: Participants] — University of Pennsylvania cytokine release syndrome (CRS) Grading System known as Penn Class defines class 3 as hypoxia requiring supplemental oxygen [nasal cannula oxygen, high-flow oxygen, continuous positive airway pressure (CPAP), or bilevel positive airway pressure (BiPAP)] and class 4 as requiring mechanical ventilation.
  Participants
    Penn Class 3 | 4 | 4 | 8
    Penn Class 4 | 6 | 6 | 12
Previous or Concomitant Therapy [Count of Participants; unit: Participants]
  Glucocorticoids | 9 | 10 | 19
  Convalescent Plasma | 2 | 7 | 9
  Remdesivir | 3 | 8 | 11
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 3 | 3 | 6
  Hypertension | 5 | 5 | 10
  Obesity | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein (CRP) Levels at Baseline and Day 14
Description: Defined as decreasing the CRP level from baseline to study day 14
Time Frame: Baseline and at Day 14
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | 1 - TPE Alone | 2 - TPE Plus Ruxolitinib
Number analyzed (Participants) | 10 | 10
mg/L
  CRP Baseline | 75.45 [41.75 to 147.9] | 59.8 [49.025 to 101.6]
  CRP Day 14 | 41.9 [17.9 to 156.2] | 38.7 [8.6 to 103.8]

2. Primary Outcome: Cytokine Levels at Baseline and Day 14
Description: Defined as decreasing the interleukin (IL) IL-6 and IL-10 load and the tumor necrosis factor (TNF) load from baseline to study day 14
Time Frame: Baseline and at Day 14
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | 1 - TPE Alone | 2 - TPE Plus Ruxolitinib
Number analyzed (Participants) | 10 | 10
pg/ml
  IL-6 Baseline | 41.32 [9.79 to 67.25] | 14.22 [7.02 to 42.07]
  IL-6 Day 14 | 14.8 [5.8 to 53.88] | 18.72 [7.4 to 31.92]
  IL-10 Baseline | 8.06 [6.22 to 20.81] | 5.6 [4.67 to 6.84]
  IL-10 Day 14 | 2 [0.56 to 3.16] | 3.16 [2.64 to 3.2]
  TNF Baseline | 10.66 [7.38 to 11.3] | 7.06 [5.02 to 10.5]
  TNF Day 14 | 9.96 [9.28 to 13.64] | 7 [5.32 to 7.56]

ADVERSE EVENTS:
Time Frame: Adverse event data collected from date of consent through study day 28
Description: As this was a hospitalized, critically ill patient population, adverse events in this study were defined as events deemed by the investigators to be related to study treatment (TPE and / or ruxolitinib). Adverse events occurring in greater than 5% of patients were reported. All serious adverse events (SAEs) were collected and reported. Patients were assessed daily by the critical care service study investigators.
Arm/Group | 1 - TPE Alone | 2 - TPE Plus Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 1/10 | 2/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - TPE Alone (N=10) | 2 - TPE Plus Ruxolitinib (N=10)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — COVID-19 related myocardial infarction
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — acute respiratory failure secondary to COVID-19
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — acute respiratory failure secondary to enterococcus bacteremia, methicillin-resistant staphylococcus aureus (MRSA)

LIMITATIONS AND CAVEATS:
Pilot study with small sample size. The imbalance between cohorts with respect to previous or concomitant therapy reflects the greater adoption of convalescent plasma and antiviral medication over the time span of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04374149/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT04374149/ICF_001.pdf